CLINICAL TRIAL: NCT04090879
Title: Low Nicotine Content Cigarettes in Vulnerable Populations: Affective Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH); University of Vermont (Other)
Responsible Party: Principal Investigator, Jennifer Tidey, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CHRMS19-0129; U54DA036114-06 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use Disorder
Keywords: Biomarkers of Exposure; Compensatory Smoking; Nicotine Dependence; Reduced Nicotine Cigarettes; Affective Disorders; Tobacco Withdrawal; Vulnerable Populations; E-Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Mood Disorders; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Randomized parallel groups research design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind dosing of tobacco cigarette nicotine levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RC 1 only (Experimental): Research Cigarettes #1
  Interventions: Other: Either normal nicotine content cigarettes (15.8mg/g) or reduced nicotine content cigarettes (0.4mg/g)
- RC 2 only (Experimental): Research Cigarettes #2
  Interventions: Other: Either normal nicotine content cigarettes (15.8mg/g) or reduced nicotine content cigarettes (0.4mg/g)
- RC 2 + EC 1 (Experimental): Research Cigarettes #2 plus E-cigarettes #1 (participants receive tobacco flavor only)
  Interventions: Other: Either normal nicotine content cigarettes (15.8mg/g) or reduced nicotine content cigarettes (0.4mg/g); Other: E-Cigarettes
- RC 2 + EC 2 (Experimental): Research Cigarettes #2 plus E-cigarettes #2 (participants can choose among varying flavors)
  Interventions: Other: Either normal nicotine content cigarettes (15.8mg/g) or reduced nicotine content cigarettes (0.4mg/g); Other: E-Cigarettes

INTERVENTIONS:
Other: Either normal nicotine content cigarettes (15.8mg/g) or reduced nicotine content cigarettes (0.4mg/g) — 1) Altering the nicotine content of the tobacco research cigarette
Other: E-Cigarettes — 1) Altering the availability of e-cigarettes; 2) Altering option to personalize the e-liquid in the e-cig condition
  Arms: RC 2 + EC 1; RC 2 + EC 2

SUMMARY:
While the prevalence of smoking in the United States general population has declined over the past 50 years, there has been little to no decline among people with mental health conditions. Affective Disorders (ADs) are the most common mental health conditions in the US, and over 40% of people with ADs are current smokers. A national policy of reducing the nicotine content of cigarettes has the potential to reduce tobacco use, dependence, and related adverse health outcomes. Controlled trials in psychiatrically-stable smokers have shown that reducing the nicotine content in cigarettes can reduce cigarettes per day (CPD), dependence and tobacco toxicant exposure, with few adverse consequences.

The goal of the proposed trial is to experimentally model whether increasing the availability and appeal of an alternative, non-combusted source of nicotine (e-cigarettes) moderates the effect of altering the nicotine in cigarettes in smokers with ADs. Additionally, investigators will test whether allowing participants to personalize the flavor of the e-liquid alters any moderating effects their availability may have on tobacco cigarette smoking.

Daily smokers with current ADs will be recruited at Brown University and the University of Vermont.

Investigators will study two research cigarettes referred to here as Research Cigarette 1 (RC1) and Research Cigarette 2 (RC2). One of these cigarettes will be a normal nicotine content cigarette and the other will be a reduced nicotine content cigarette. Investigators will study two e-cigarette conditions referred to here as E-Cigarette Condition 1 (EC1) and E-Cigarette Condition 2 (EC2). Both e-cigarette conditions will involve the same commercially available devices and same nicotine-containing e-liquid, but in one condition that e-liquid will be available only in tobacco flavor while in the other condition that e-liquid will be available in multiple flavors from which participants can choose based on personal taste preference. Participants will be assigned to one of the following four study conditions: (1) RC1 only; (2) RC2 only; (3) RC2 + EC1; (4) RC2 + EC2.

Participants will be asked to use only their assigned study products for 16 weeks. Outcome measures include total CPD, cigarette demand assessed by behavioral economics-based purchase tasks, craving, withdrawal, psychiatric symptoms, breath carbon monoxide (CO), biomarkers of tobacco toxicant exposure, brain function and structure, and airway inflammation (fractional nitric oxide concentration in exhaled breath [FeNO]).

ELIGIBILITY:
Inclusion Criteria

* Between 21 years and 70 years old
* Must have current diagnosis of an Affective Disorder.

Exclusion Criteria

* Being without an Affective Disorder
* Younger than 21 years old
* Older than 70 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W Tidey, Ph.D., Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Brown University, Providence, Rhode Island
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Higgins ST, Sigmon SC, Tidey JW, Heil SH, Gaalema DE, Lee DC, DeSarno MJ, Klemperer EM, Menson KE, Cioe PA, Plucinski S, Wiley RC, Orr E. Reduced Nicotine Cigarettes and E-Cigarettes in High-Risk Populations: 3 Randomized Clinical Trials. JAMA Netw Open. 2024 Sep 3;7(9):e2431731. doi: 10.1001/jamanetworkopen.2024.31731. PMID 39240566

RESULTS

PARTICIPANT FLOW:
Groups:
- RC 1 Only: Research Cigarettes #1
  Participants in this group were randomized to receive normal nicotine content cigarettes (15.8mg/g) only, and e-cigarettes were not available. This condition of the intervention applied to these participants throughout all timepoints of the study
  1. Altering the nicotine content of the tobacco research cigarette
  2. Altering the availability of e-cigarettes
- RC 2 Only: Research Cigarettes #2
  Participants in this group were randomized to receive reduced nicotine content cigarettes (0.4mg/g) only, and e-cigarettes were not available. This condition of the intervention applied to these participants throughout all timepoints of the study
  1. Altering the nicotine content of the tobacco research cigarette
  2. Altering the availability of e-cigarettes
- RC 2 + EC 1: Research Cigarettes #2 plus E-cigarettes #1 (participants receive tobacco flavor only)
  Participants in this group were randomized to receive reduced nicotine content cigarettes (0.4mg/g) only, and tobacco flavor e-cigarettes only. This condition of the intervention applied to these participants throughout all timepoints of the study
  1. Altering the nicotine content of the tobacco research cigarette
  2. Altering the availability of e-cigarettes
  3. Altering option to personalize the e-liquid in the e-cig condition
- RC 2 + EC 2: Research Cigarettes #2 plus E-cigarettes #2 (participants can choose among varying flavors)
  Participants in this group were randomized to receive reduced nicotine content cigarettes (0.4mg/g) only, and were given availability to a variety of flavors, and thus were able to select preferred flavor. This condition of the intervention applied to these participants throughout all timepoints of the study
  1. Altering the nicotine content of the tobacco research cigarette
  2. Altering the availability of e-cigarettes
  3. Altering option to personalize the e-liquid in the e-cig condition
Period: Overall Study
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
Started | 83 | 85 | 74 | 84
Completed | 67 | 66 | 57 | 70
Not Completed | 16 | 19 | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2 | Total
Number analyzed (Participants) | 83 | 85 | 74 | 84 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.77 (10.98) | 39.85 (9.28) | 41.51 (12.39) | 39.38 (10.59) | 40.09 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 69 | 50 | 59 | 243
  Male | 18 | 16 | 24 | 25 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Latino | 9 | 6 | 9 | 9 | 33
  Latino | 4 | 3 | 3 | 2 | 12
  White, non-Latino | 66 | 68 | 60 | 68 | 262
  Non-Latino other or multiracial | 4 | 8 | 2 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 83 | 85 | 74 | 84 | 326
Population [Count of Participants; unit: Participants]
  Females with lower educational level | 20 | 23 | 16 | 21 | 80
  OUD | 19 | 19 | 17 | 19 | 74
  Affective disorders | 44 | 43 | 41 | 44 | 172
Educational level [Count of Participants; unit: Participants]
  <High school | 9 | 4 | 3 | 14 | 30
  High school graduate, equivalency, or some college | 51 | 57 | 46 | 47 | 201
  Associate's degree | 8 | 11 | 13 | 11 | 43
  ≥College graduate | 15 | 13 | 12 | 12 | 52
Marital status [Count of Participants; unit: Participants]
  Married | 8 | 15 | 17 | 11 | 51
  Never married | 49 | 47 | 36 | 48 | 180
  Divorced, separated, or widowed | 26 | 23 | 21 | 25 | 95
Primarily smokes mentholated cigarettes [Count of Participants; unit: Participants] | 32 | 35 | 31 | 33 | 131
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] | 16.42 (8.02) | 18.44 (9.47) | 17.86 (9.11) | 16.90 (8.85) | 17.40 (8.87)
Urine cotinine level [Mean (Standard Deviation); unit: ng/mL] | 4499.25 (3120.20) | 5235.67 (3251.28) | 5156.57 (4150.44) | 5293.33 (3799.45) | 5043.55 (3680.12)
Breath CO level [Mean (Standard Deviation); unit: ppm] | 20.90 (14.02) | 19.30 (12.39) | 21.03 (13.38) | 20.66 (13.44) | 20.46 (13.28)
Age started smoking regularly [Mean (Standard Deviation); unit: years] | 16.61 (3.97) | 15.92 (3.91) | 16.24 (3.84) | 16.79 (5.15) | 16.39 (4.26)
FTND total score [Mean (Standard Deviation); unit: scores on a scale] — Fagerstrom Test for Nicotine Dependence
  In scoring the Fagerstrom Test for Nicotine Dependence, the three yes/no items are scored 0 (no) and 1 (yes). Two of the three multiple-choice items are scored from 0 to 3, with the third multiple choice item being scored from 0 to 1.
  The items are summed to yield a total score of 0-10.
  Classification of dependence based on total score:
  0-2 Very low 3-4 Low 5 Moderate 6-7 High 8-10 Very high
  scores on a scale | 5.12 (2.24) | 5.31 (2.20) | 5.26 (2.31) | 4.70 (2.07) | 5.09 (2.21)
Used other tobacco products, past 30 days [Count of Participants; unit: Participants] | 5 | 4 | 5 | 9 | 23
Used e-cigarettes, past 30 days [Count of Participants; unit: Participants] | 13 | 11 | 5 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Day
Description: Cigarettes per day will be assessed for use of cigarettes with different nicotine content.
Time Frame: 16 weeks
Population: Participants who completed week 16 of study
Measure: Least Squares Mean (Standard Error); unit: cigarettes per day
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
Number analyzed (Participants) | 67 | 66 | 57 | 70
cigarettes per day | 22.54 (1.59) | 14.32 (1.32) | 11.76 (1.18) | 7.63 (0.90)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/85 | 1/74 | 0/84
Serious Adverse Events (participants affected / at risk) | 9/83 | 4/85 | 4/74 | 2/84
Other Adverse Events (participants affected / at risk) | 71/83 | 74/85 | 62/74 | 72/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC 1 Only (N=83) | RC 2 Only (N=85) | RC 2 + EC 1 (N=74) | RC 2 + EC 2 (N=84)
Psychiatric disorders - Other (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy, puerperium, and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC 1 Only (N=83) | RC 2 Only (N=85) | RC 2 + EC 1 (N=74) | RC 2 + EC 2 (N=84)
OASIS Score Increase (Psychiatric disorders) | 32 (51) | 31 (43) | 31 (42) | 31 (40)
BDI Category Increase (Psychiatric disorders) | 29 (51) | 29 (40) | 26 (34) | 25 (41)
Psychiatric disorders (Psychiatric disorders) | 27 (53) | 28 (43) | 19 (27) | 24 (37)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 23 (38) | 27 (44) | 18 (40) | 18 (35)
General disorders and administration (General disorders) | 18 (25) | 24 (27) | 16 (20) | 22 (27)
Infections and infestations (Infections and infestations) | 16 (17) | 23 (24) | 8 (11) | 10 (13)
Nervous system disorders (Nervous system disorders) | 7 (8) | 18 (23) | 15 (19) | 10 (11)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (14) | 17 (25) | 14 (20) | 17 (23)
Vascular disorders (Vascular disorders) | 10 (13) | 13 (15) | 8 (10) | 16 (30)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 (14) | 16 (16) | 7 (7) | 12 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 (7) | 4 (7) | 4 (4) | 5 (8)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 3 (3) | 5 (5) | 4 (4)
Cardiac disorders (Cardiac disorders) | 4 (6) | 2 (4) | 3 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT04090879/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT04090879/ICF_001.pdf